CLINICAL TRIAL: NCT04530071
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1/2a, Multi-center Clinical Trial for Evaluation of Safety, Tolerability, and Efficacy of CordSTEM-DD in Patients With Chronic Low Back Pain Due to Lumbar Intervertebral Disc Degeneration
Brief Title: Evaluation of Safety, Tolerability, and Efficacy of CordSTEM-DD in Patients With Chronic Low Back Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHABiotech CO., Ltd (Industry)
Collaborators: Seoul CRO Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CHA-CDD-101
Record Dates: First submitted 2020-08-19; First posted 2020-08-28 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Chronic Low-back Pain; Disc Degeneration
Keywords: Stem Cell therapy; Cell therapy; Disc Degeneration; Back pain
MeSH Terms: conditions — Intervertebral Disc Degeneration; Back Pain

STUDY DESIGN:
Intervention Model Description: Double-blinding will be used to prevent subjective biases of the subjects and the investigator from affecting the study results.
  Subject assignment group will be disclosed only to the unblinded sub-investigator or unblinded study coordinator and unblinded investigator designated as a person responsible for IP management and procedures.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CordSTEM-DD(0.7x10^7 cells) (Experimental): HA+saline+CordSTEM-DD(0.7x10^7 cells)
  Interventions: Biological: CordSTEM-DD (0.7 x 10^7 cells)
- CordSTEM-DD(2.1x10^7 cells) (Experimental): HA+saline+CordSTEM-DD(2.1x10^7 cells)
  Interventions: Biological: CordSTEM-DD (2.1 x 10^7 cells)
- Control group (Placebo Comparator): HA + saline + placebo comparator
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CordSTEM-DD (0.7 x 10^7 cells) — CordSTEM-DD (0.7 x 10^7 cells)
  Arms: CordSTEM-DD(0.7x10^7 cells)
Biological: CordSTEM-DD (2.1 x 10^7 cells) — CordSTEM-DD (2.1 x 10^7 cells)
  Arms: CordSTEM-DD(2.1x10^7 cells)
Biological: Placebo — HA + saline + placebo comparator
  Arms: Control group

SUMMARY:
The purpose of this clinical study is to evaluate the safety, tolerability, and efficacy of CordSTEM-DD, an allogeneic umbilical cord-derived mesenchymal stem cell, as a cell-therapeutic drug in patients with chronic low back pain due to lumbar intervertebral disc degeneration.

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, placebo-controlled, single-dose, phase 1/2a, multi-center study to evaluate the safety, tolerability, and efficacy of the treatment with CordSTEM-DD, an allogeneic umbilical cord-derived mesenchymal stem cell, in patients with chronic low back pain due to lumbar intervertebral disc degeneration.

During the study period, subjects will have a total of 8 visits: Week 2, Month 1, Month 3, Month 6, Month 9 and Month 12, in addition to screening and baseline visits.

The primary objective will include assessment of safety and tolerability for 12 months after the administration of the study drug. Safety will be assessed based on the results of adverse events, confirmation of malignancy, all deaths, laboratory tests, and physical examinations/vital signs. As the secondary objective, efficacy will be assessed by identifying the Visual Analogue Scale (VAS), Oswestry Disability Index (ODI ), treatment success rate, The 36-Item Short Form Health Survey (SF-36) score, and change on lumbar MRI.

This clinical study consists of Stage I and Stage II, and the composition of the study group and the control group in each stage and the number of subjects to be enrolled are as follows:

[Stage I]

* Group 1 (3 subjects): Hyaluronic Acid (HA) + saline + study drug (0.7 × 10^7 cells CordSTEM-DD)
* Group 2 (3 subjects): HA + saline + study drug (2.1 × 10^7 cells CordSTEM-DD) [Stage II] After confirming the safety of the administered dose of the investigational product in Stage I, an additional 30 subjects will be recruited and randomized.
* Control group (10 subjects): HA + saline + comparator
* Group 1 (10 subjects): HA + saline + study drug (0.7 × 10^7 cells CordSTEM-DD)
* Group 2 (10 subjects): HA + saline + study drug (2.1 × 10^7 cells CordSTEM-DD)

ELIGIBILITY:
Inclusion Criteria:

1. Male and females aged ≥ 19 years and < 70 years
2. Have low back or hip pain that has lasted ≥ 6 months at the time of screening and do not respond to conservative therapy* given for ≥ 3 months

   * Conservative therapy: Rest at an early stage, drug treatment (e.g., anti-inflammatory drugs, analgesics, anesthetics, narcotic analgesics, muscle relaxants), massage, acupuncture, chiropractic treatment, posture correction, home lumbar exercise programs, etc.
3. The Oswestry Disability Index (ODI) of 30% or greater and below 90% at screening
4. The Visual Analogue Scale (VAS) score for pain in the lumbar spine of ≥ 40 mm and ≤ 90 mm in the last 3 months prior to screening
5. The magnetic resonance imaging (MRI) grade 3 to 6 between lumbar vertebra 1 and sacral vertebra 1 according to the modified Pfirrmann classification method at screening
6. One pain-causing degenerative lumbar disc identified at screening. However, degenerative lumbar discs causing pain are identified by discography.
7. Those who provide written consent to comply with the precautions after they or their representatives voluntarily decide to participate subsequent to listening to a detailed explanation of this clinical study and understanding it completely

Exclusion Criteria:

1. Body mass index (BMI) of 30 ㎏/m2 or greater
2. Those who require surgery because they have symptoms of nerve compression due to severe lumbar spinal stenosis or lumbar herniated nucleus pulposus
3. Those with spinal instability, spondylitis, or vertebral fractures
4. Severe degenerative changes in the intervertebral disc leading to a 30% or more decrease in the height of the intervertebral disc
5. Those who have modic type 3 changes on MRI
6. Those with severe osteoporosis

   * An average T score of -2.5 or less in the lumbar bone density test (DEXA, Dual-Energy X-ray Absorptiometry)
7. Those who have undergone procedures (electrocoagulation of the intervertebral disc, etc.) and surgery such as discectomy on the disc to be administered with the investigational product However, in the case of electrocoagulation, enrollment is allowed if the procedure was performed 3 months prior to the administration of the investigational product on the annulus fibrosus, not on the nucleus pulposus.
8. Those who took at least 75 mg/day of morphine equivalent dose (MED) during the screening period
9. Those who have full-thickness annular tears (modified Dallas diagram scale grade 5) at index level when a contrast medium is administered to annulus fibrosus (AF)
10. Those with clinically significant neuralgia (e.g., chronic radiculopathy) or neuropathy
11. Those with clinically significant sacroiliac joint pain
12. Those who have compressive pathology due to stenosis or disc extrusion confirmed by MRI, and have clinical symptoms of leg pain with VAS of 40 mm or more, or a neurological deficit confirmed in a neurological examination
13. Those with intermittent neurogenic claudication due to central vertebral canal stenosis
14. Those with lumbar spondylitis or ankylosing spondylitis caused by autoimmune diseases, etc.
15. Those with facet joint pain confirmed through a diagnostic medical branch block
16. Those who have received an injection of a drug containing steroids into the disc, except for the following drugs, within 3 weeks of the administration of the investigational product (1) Contrast medium (discography or other diagnostic injection) (2) Non-steroidal anti-inflammatory drugs (NSAIDs) (3) Nerve-blocking local anesthetics: e.g., lidocaine, bupivacaine (4) Antibiotics (5) Normal saline (saline)
17. Those who have a history of malignancy within 5 years of screening
18. Those taking systemic immunosuppressants
19. Those who have received biological treatments such as proteins and antibody treatments for the treatment of degenerative disc disease (DDD)
20. Those who have received intravertebral cell-therapeutic drugs or platelet rich plasma (PRP) therapy (However, enrollment is allowed if stem cell therapy was administered by a route other than the intervertebral disc and ≥ 5 years have passed)
21. Those who may affect this clinical study due to serious medical disease [uncontrolled hypertension, uncontrolled diabetes mellitus, uncontrolled active infection or tuberculosis, cirrhosis of the liver, kidney failure, tumors, etc.]
22. Those with a history of allergy to protein products (bovine serum), antibiotics (gentamicin), DMSO, and hyaluronic acid (HA) required for the manufacture of cell-therapeutic drugs
23. Those who have a psychiatric history or are being treated, and the investigator determines that it is difficult to proceed with the clinical study
24. Those who exceed 30 points on the Beck Depression Inventory (BDI)
25. Those who cannot understand the purpose, method, etc. of this clinical study due to drug or alcohol addiction
26. Those who participated in other clinical studies within 6 months prior to participation in this clinical study
27. Pregnant or breastfeeding women
28. Male or female patients of childbearing potential who do not agree to use medically acceptable methods of contraception* during the clinical study period

    * Medically acceptable methods of contraception: Condoms, oral contraceptives for at least 3 months, injectable contraceptive procedure performed 3 months ago, use of injectable or implantable contraceptives, intrauterine contraceptive devices, etc.
29. Those who are ineligible for participation in the clinical study in the judgment of the principal investigator or sub-investigator due to other ethical reasons or reasons that may affect the results of the clinical study

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events during the study period | 28 days on Stage 1
Number of treatment emergent adverse events during the study period | 12 months on Stage 2

CONTACTS AND LOCATIONS:
Overall Officials: In-Bo Han, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA Bundand Medical Center, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No